CLINICAL TRIAL: NCT04120974
Title: The Role of Proper Insulin Injection Technique in the Treatment of Diabetes
Brief Title: The Role of Proper Insulin Injection Technique in the Treatment of Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBC-19INJCTRU; BD-4MM (Other: Becton Dickinson)
Record Dates: First submitted 2019-10-04; First posted 2019-10-09 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Lipohypertrophy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optimal insulin injection (Experimental): Study subjects will receive personal training from the Investigator on how to optimally inject insulin to treat their Diabetes Mellitus. In addition, each subject receives instruction how to use a web-based platform with online video training modules on optimal injection technique.
  Interventions: Behavioral: Optimal insulin injection

INTERVENTIONS:
Behavioral: Optimal insulin injection — subjects receive training in optimal injection technique.

SUMMARY:
This is a prospective, post-marketing, single-arm clinical investigation on the effects of optimal insulin injection technique, in conjunction with the use of disposable Becton Dickinson (BD) Micro-Fine Plus 32G pen needles, by Type I and Type II Diabetes Mellitus patients, with or without lipohypertrophy, on clinical outcomes like HbA1c and hypoglycemic events, as well as changes in insulin Total Daily Dose (TDD) and patient's Quality of Life (QoL). During this study, each subject will be trained in the optimal insulin injection technique by personal training as well as by following online video training modules on a specific web-based platform.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or type 2 diabetes mellitus;
2. At least 1 year of experience with insulin self-administration;
3. Use of insulin pen for insulin injections.
4. HbA1c > 7.5 % measured at study entry or maximally 30 days prior to screening.
5. BMI below 40 kg/m2 at study entry.
6. Daily self-control of blood glucose level;
7. Access to the internet for watching video lessons.
8. Only outpatients are eligible for the study.
9. Availability of signed informed consent of the patient for inclusion in the study.

Exclusion Criteria:

1. Pregnant women or women planning to become pregnant during the time of study, breastfeeding women;
2. Subjects using an insulin pump;
3. Those using treatment with a Glucagon-Like Peptide (GLP)-1 receptor agonists alone;
4. Subjects not fluent in Russian (reading and writing).
5. Patients at high risk for ketoacidosis and/or hyperglycemia.
6. Psychic, physical or any other reasons hampering patient participation in the study (based on the reasonable opinion of the physician-investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Mayorov, MD, Principal Investigator — National Medical Research Center of Endocrinology (ENC)
Locations (4):
- Russia (4):
  - National Medical Research Center of Endocrinology (ENC), Moscow
  - Moscow Regional Research Clinical Institute (MONIKI), Moscow
  - Endocrinological Dispensary of the Moscow Department of Health (DZM), Moscow
  - State Healthcare Institution "Sverdlovsk Regional Clinical Hospital No. 1" (EKB), Yekaterinburg

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Optimal Insulin Injection Technique: Patients with Type I or Type II Diabetes Mellitus with an HbA1c value >7.5% and at least 1 year experience with insulin self-administration were enrolled in this study. Patients were re-trained in the correct technique of insulin injection and received access to video training modules.
Period: Overall Study
Arm/Group | Optimal Insulin Injection Technique
Started | 90
Completed | 82
Not Completed | 8
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: Only the participants who completed the study have been analyzed and are reported on. 90 Participants included, but 82 completed the study.
Arm/Group | Optimal Insulin Injection Technique
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 82
BMI, average [Mean (Standard Deviation); unit: kg/m^2] | 26.7 (5.1)
Baseline HbA1c (%), average [Mean (Standard Deviation); unit: % of glycated hemoglobin] | 9.2 (1.4)
Diabetes Type: Type I, Type II [Count of Participants; unit: Participants]
  Type I Diabetes Mellitus | 57
  Type II Diabetes Mellitus | 25
Insulin therapy duration, average (years) [Mean (Standard Deviation); unit: years] | 13.2 (11.4)
Baseline Lipohypertrophy: Yes, No [Count of Participants; unit: Participants]
  Lipohypertrophy present | 46
  Lipohypertrophy absent | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycemic Control
Description: Change in HbA1c for subjects from Baseline to 6 months; expressed as theHbA1c% levels at Baseline and 6-months
Time Frame: up to 6 months
Population: Only participants who completed the study have been analyzed
Measure: Mean (Standard Deviation); unit: % of glycated hemoglobin
Arm/Group | Optimal Insulin Injection Technique
Number analyzed (Participants) | 82
% of glycated hemoglobin
  HbA1c at Baseline | 8.99 (1.37)
  HbA1c at 6-months follow up | 8.20 (1.10)

2. Secondary Outcome: Change in Insulin Total Daily Dose (TDD)
Description: Change in Insulin TDD for subjects from Baseline to 3 and 6 months; expressed as the Total Units at Baseline, 3-months and 6-months follow up
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Optimal Insulin Injection Technique
Number analyzed (Participants) | 82
units
  TDD Insulin at Baseline | 49.5 (24.1)
  TDD Insulin at 3-months follow up | 49 (24.1)
  TDD Insulin at 6-months follow up | 51.2 (26.7)

3. Secondary Outcome: Incidence of Hypoglycemic Events
Description: Incidence rate of hypoglycemic events in the 2-week period at study start (Baseline), a 2-week period approximately 3 months after Baseline, and during a 2 week period around 6 months follow up, expressed in per person-year
Time Frame: up to 6 months
Population: Data are expressed as overall (all participants) and split per type of Diabetes (Type I or Type II)
Measure: Number; unit: events per person-year
Arm/Group | Optimal Insulin Injection Technique
Number analyzed (Participants) | 82
events per person-year
  Incidence of hypoglycemic events at Baseline (overall) | 56.15
  Incidence of hypoglycemic events at 3-months follow up (overall) | 36.35
  Incidence of hypoglycemic events at 6-months follow up (overall) | 32.28
  Incidence of hypoglycemic events at Baseline (Type I DM): number analyzed (Participants) | 57
  Incidence of hypoglycemic events at Baseline (Type I DM) | 74.42
  Incidence of hypoglycemic events at 3-months follow up (Type I DM): number analyzed (Participants) | 57
  Incidence of hypoglycemic events at 3-months follow up (Type I DM) | 52.66
  Incidence of hypoglycemic events at 6-months follow up (Type I DM): number analyzed (Participants) | 57
  Incidence of hypoglycemic events at 6-months follow up (Type I DM) | 42.62
  Incidence of hypoglycemic events at Baseline (Type II DM): number analyzed (Participants) | 25
  Incidence of hypoglycemic events at Baseline (Type II DM) | 21.04
  Incidence of hypoglycemic events at 3-months follow up (Type II DM): number analyzed (Participants) | 25
  Incidence of hypoglycemic events at 3-months follow up (Type II DM) | 7.43
  Incidence of hypoglycemic events at 6-months follow-up (Type II DM): number analyzed (Participants) | 25
  Incidence of hypoglycemic events at 6-months follow-up (Type II DM) | 11.82

4. Secondary Outcome: Change in Blood Glucose Levels
Description: Change in average Blood Glucose Levels (measured by a Blood Glucose Meter) of the first 2 weeks after enrolment (Baseline), compared to the average Blood Glucose Levels during 2 weeks around 3 month and the average of 2 weeks Blood Glucose Levels around 6 months; expressed as mmol/L
Time Frame: up to 6 months
Population: Not all participants had BGM data available, this is the reason the number of analyzed participants deviates from the total number analyzed in the study.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Optimal Insulin Injection Technique
Number analyzed (Participants) | 72
mmol/L
  24-hour blood glucose average during a two-week period at Baseline | 10.28 (3.04)
  24-hour blood glucose average during a two-week period at 3-months follow up: number analyzed (Participants) | 69
  24-hour blood glucose average during a two-week period at 3-months follow up | 11.03 (3.13)
  24-hour blood glucose average during a two-week period at 6-months follow up: number analyzed (Participants) | 66
  24-hour blood glucose average during a two-week period at 6-months follow up | 11.03 (3.45)

5. Other Pre Specified Outcome: Effect on Quality of Life
Description: In the EQ-5D-35L the 5 dimensions are described by 3 problem levels corresponding to subject response choices.
  A quality of life score (Health State Index Score) is obtained according to the answers to the questionnaires. The scale runs from 0 to 1, higher scores mean a better quality of life.
  Quality of Life scores will be reported at Baseline and at 6 months;
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Optimal Insulin Injection Technique
Number analyzed (Participants) | 82
score on a scale
  Health State Index Score at Baseline | 0.76 (0.21)
  Health State Index Score at 6-months follow up | 0.78 (0.24)

6. Other Pre Specified Outcome: Change in Needle Re-use
Description: Rate of needle re-use by self-reporting, expressed as number of participants reporting single-use needles at Baseline and after 3- and 6 months.
  Study participants were queried on their injection technique during study follow up visits and it was documented if they responded the use of a new needle for each insulin injection (single-use needles).
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Optimal Insulin Injection Technique
Number analyzed (Participants) | 82
Participants
  Single needle use at Baseline | 4
  Single needle use at 3-month follow up | 66
  Single needle use at 6-month follow- up | 73

7. Other Pre Specified Outcome: Effect on Lipohypertrophy Areas
Description: Sub-group: for subjects with lipohypertrophy areas at enrolment, change in lipohypertrophy size (length and width) from Baseline to 6 months At Baseline, lipohypertrophy areas caused by repeated insulin injections at the same injection location, were measured. These areas were measured again during the 3-month and 6-month follow up visits.
Time Frame: up to 6 months
Population: Only participants with lipohypertrophy at Baseline were included in this analysis
Measure: Geometric Mean (Standard Deviation); unit: cm
Arm/Group | Optimal Insulin Injection Technique
Number analyzed (Participants) | 46
cm
  Length lipohypertrophy area at Baseline | 4.13 (2.63)
  Length lipohypertrophy area at 3-months follow up | 3.61 (2.16)
  Length lipohypertrophy area at 6-months follow up | 3.18 (1.80)
  Width lipohypertrophy area at Baseline | 3.69 (2.47)
  Width lipohypertrophy area at 3-months follow up | 3.17 (1.88)
  Width lipohypertrophy area at 6-months follow up | 3.07 (1.92)

8. Other Pre Specified Outcome: Effect on Behaviour: Injection in Lipohypertrophy Areas
Description: Sub-group: for subjects with lipohypertrophy areas at enrolment, change in injection into lipohypertrophy areas from Baseline to 6 months Study participants were queried on their injection technique during study baseline and follow up visits and it was documented if they responded if they inject insulin at a location with lipohypertrophy or at a different location for each injection (rotating).
Time Frame: up to 6 months
Population: Only participants with lipohypertrophy at Baseline were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Optimal Insulin Injection Technique
Number analyzed (Participants) | 46
Participants
  Injection in lipohypertrophy area at Baseline | 40
  Injection in lipohypertrophy area at 3-months follow up | 1
  Injection in lipohypertrophy area at 6-months follow up | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from study enrollment until End of Study (between Baseline and approximately 6-months follow up)
Description: Adverse Event collection was systematically collected by study site staff during on-site and telephone follow-up visits. A Clinical Research Associate has conducted a 100% source data verification and reviewed patient medical charts to ensure all Adverse Events were captured in the Case Report Forms.
Arm/Group | Optimal Insulin Injection Technique
All-Cause Mortality (participants affected / at risk) | 1/90
Serious Adverse Events (participants affected / at risk) | 4/90
Other Adverse Events (participants affected / at risk) | 5/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimal Insulin Injection Technique (N=90)
COVID-19 (Infections and infestations) | 1 (1) — COVID-19
COVID-19 pneumonia (Infections and infestations) | 1 (1) — COVID-19 and bilateral polysegmental pneumonia due to COVID-19.
Death (General disorders) | 1 (1) — The cause is not clear, the statement in the documents mentions "other unspecified causes of death".
Coronary artery disease (Cardiac disorders) | 1 (1) — Planned hospitalization for coronography due to coronary heart disease.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimal Insulin Injection Technique (N=90)
Visual impairment (Eye disorders) | 1 (1) — Vision problem induced by Diabetes Mellitus
Hypotension (Vascular disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) — Foot ulcer and necessity to wear foot cast
Nasopharyngitis (Infections and infestations) | 1 (1) — Acute respiratory infection - rhinopharyngitis
Respiratory tract infection viral (Infections and infestations) | 1 (1) — Acute respiratory viral infection (clinically COVID-19 was probable, but was not confirmed)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT04120974/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT04120974/SAP_001.pdf